CLINICAL TRIAL: NCT01896843
Title: Evaluation of [11C]FPEB, [18C]FPEB, and [11C]SP203 To Image mGluR5 Receptors In Brain
Brief Title: Evaluation of Two Radioactive Chemicals to Image mGluR5 Receptors in Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130166; 13-M-0166
Record Dates: First submitted 2013-07-02; First posted 2013-07-11 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2017-01-11

CONDITIONS: mGluR5 Receptors
Keywords: Positron Emission Tomography (PET); Metabotropic Glutamate Receptors

INTERVENTIONS:
Drug: STX107

SUMMARY:
Background:

- A small brain protein called the metabotropic glutamate receptor subtype 5 (mGluR5) may affect several brain diseases such as autism and depression. Researchers will use 2 radioactive chemicals ([11C]SP203 and [11C]FPEB) and a research drug (STX107) that can attach to the receptor, to figure out the best way to use positron emission tomography (PET) to see the mGluR5 receptor. They will use scans to monitor where the radioactivity goes.

Objectives:

- To find the best way to image the mGluR5 receptor in the brain.

Eligibility:

- Healthy volunteers ages 18 to 55.

Design:

* All participants will be screened with a medical exam at visit 1. In later visits, they may have a PET scan, when two small tubes are placed under the skin and they lie down in a scanner. They may have an MRI scan, when they lie down in a scanner.
* Part 1 participants will have 2 more visits. They will have a PET brain scan using [11C]FPEB and will have blood drawn. Then they will have an MRI brain scan.
* Part 2 participants will have 1 more visit, with a whole body PET scan using [11C]FPEB and blood drawn.
* Part 3 participants will have 4 more visits, including 1 overnight stay at a hospital. Over all the visits, they will have 4 PET scans and 1 MRI brain scan. They will receive the research drug and injections of both chemicals. Blood will be drawn during the scans.

DETAILED DESCRIPTION:
Objective:

Multiple PET ligands exist for imaging metabotropic glutamate receptor subtype 5 (mGluR5). The selection of best PET ligand to image mGluR5 is necessary for a larger clinical study in patient population but choosing such a ligand is likely difficult because the radioligands are evaluated under different conditions and in different subject populations.

The purpose of this study is to determine the best PET ligand for imaging mGluR5 receptors in brain of healthy subjects. This will be accomplished by measuring mGluR5 receptor occupancy in the same subject using two PET ligands having high affinity at mGluR5 [(11)C]SP203 and [(11)C]FPEB, and using STX107, a negative allosteric modulator at mGluR5 receptors to block the radioligand brain uptake. The two radioligands were chosen among many based on the recommendation from the mGluR5 working group. Two serial PET scans using [(11)C]SP203 and [(11)C]FPEB will be performed under baseline condition on one day and under receptor blocked condition on another day. As [(11)C]FPEB has not been evaluated in humans before, we plan to acquire brain and whole-body dosimetry scans before measuring receptor occupancy.

Furthermore, we wish to compare FPEB labeled with (11)C and (18)F in the same subject -two brain PET scans using [(11)C]FPEB and [(18)F]FPEB will be done serially in the same subject on the same day. FPEB labeled with (11)C has the same structure as FPEB labeled with (18)F and is therefore expected to yield similar binding measures.

Study population:

55 healthy volunteers aged 18 to 55 years.

Design:

To characterize brain uptake and distribution of radioligand, an initial cohort of healthy volunteers (n = up to 10) will undergo brain PET scans using [(11)C]FPEB. To estimate radiation absorbed doses for [(11)C]FPEB, a cohort of healthy volunteers (n = up to 10) will undergo whole-body PET or PET/CT scans. A subsequent cohort of healthy volunteers (n = up to 15) will have two scanning sessions: a) baseline i.e., medication-free and b) blocking i.e. with medication. Each scanning session will be with two serial PET scans: [(11)C]FPEB and [(11)C]SP203 in a day (scans in morning and afternoon). The blocking session will be after administration of STX107, at which time we will also measure the concentration of STX107 in plasma. Both scanning sessions would include an arterial line and measurement of the input function of parent radioligand separated from radiometabolites as well as plasma free fraction of radioligand. We plan to study up to two doses of STX107, with three to five subjects at each dose. The blockade of brain uptake of [(11)C]FPEB and [(11)C]SP203 will be plotted as a function of the plasma concentration of STX107. A further cohort of healthy volunteers (n = up to 15) will undergo two serial brain PET scans with [(11)C]FPEB and [(18)F]FPEB in the same day (one scan in the morning, and the other in the afternoon).

Outcome measures:

The radioligands will be evaluated on three criteria:

1. Peak brain uptake. Higher uptake is better, because it provides more robust signal that can be imaged for a longer time.
2. Time-stability of distribution volume. If the measurement of receptor binding (i.e., distribution volume) is stable with increasing lengths of imaging, the result is good and consistent with the lack of radiometabolites in brain.
3. Ratio of specific to non-displaceable uptake in brain. The receptor occupancy study can be analyzed with the so-called Lassen plot to calculate non-displaceable (free radioligand plus non-specifically bound) uptake in brain. The better radioligand has the better ratio of signal to noise , which in this case is the ratio of specific to nondisplaceable uptake.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or female subjects between 18 to 55 yrs of age and able to give written informed consent.
  2. Subjects must be healthy based on medical history, physical examination and laboratory testing.

EXCLUSION CRITERIA:

1. Any past or present Axis I psychiatric disorder. Any history of alcohol or substance dependence, except nicotine dependence, within the past 6 months
2. Serious medical problems including but not limited to chronic neurological disease such as multiple sclerosis, autoimmune diseases, or serious cardiopulmonary disease.
3. Active seizure disorder, as defined as having had a seizure in the past year or being on antiepileptic medications for seizures.
4. Positive HIV test.
5. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
6. Metallic foreign bodies that would be affected by the MRI magnet or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
7. Positive urine drug screen at time of enrollment.
8. Pregnancy at time of scan (Beta-HCG will be measured in all female patients within 24 hours before start of scan and must be negative). Lactating women who are breast feeding.
9. Prescription or over-the counter medication use; psychotropic herb use (e.g., St. John s Wort).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-06-27; Primary Completion 2016-06-16 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Peak brain uptake, Time-stability of distribution volume, Ratio of specific to non-displaceable brain uptake | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ametamey SM, Treyer V, Streffer J, Wyss MT, Schmidt M, Blagoev M, Hintermann S, Auberson Y, Gasparini F, Fischer UC, Buck A. Human PET studies of metabotropic glutamate receptor subtype 5 with 11C-ABP688. J Nucl Med. 2007 Feb;48(2):247-52. PMID 17268022
- [Background] Backstrom P, Hyytia P. Ionotropic and metabotropic glutamate receptor antagonism attenuates cue-induced cocaine seeking. Neuropsychopharmacology. 2006 Apr;31(4):778-86. doi: 10.1038/sj.npp.1300845. PMID 16123768
- [Background] Bear MF, Huber KM, Warren ST. The mGluR theory of fragile X mental retardation. Trends Neurosci. 2004 Jul;27(7):370-7. doi: 10.1016/j.tins.2004.04.009. PMID 15219735